CLINICAL TRIAL: NCT02211937
Title: Relative Oral Bioavailability of 400 mg BI 44847 as Suspension Compared to 400 mg BI 44847 as Tablet and the Influence of Food (Standardised High Fat Breakfast) on the Tablet in a Single Dose, Open-label, Randomised Three-way Crossover Trial and Relative Oral Bioavailability of 40 mg BI 44847 as Solution Compared to 40 mg BI 44847 as Tablet in Healthy Male Volunteers in a Single Dose, Open-label, Randomised Two-way Crossover Trial
Brief Title: Relative Oral Bioavailability of BI 44847 as Suspension Compared to Tablet and the Influence of Food Anf of BI 44847 as Solution Compared to Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1224.2
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (5):
- Treatment A (Active Comparator): BI 44847 suspension high dose, fasted
  Interventions: Drug: BI 44847 suspension, high dose
- Treatment B (Experimental): BI 44847 tablet high dose, fasted
  Interventions: Drug: BI 44847 tablet, high dose
- Treatment C (Experimental): BI 44847 tablet high dose, fed
  Interventions: Drug: BI 44847 tablet, high dose; Other: high fat breakfast
- Treatment D (Active Comparator): BI 44847 solution low dose, fasted
  Interventions: Drug: BI 44847 solution, low dose
- Treatment E (Experimental): BI 44847 tablet low dose, fasted
  Interventions: Drug: BI 44847 tablet, low dose

INTERVENTIONS:
Drug: BI 44847 solution, low dose
  Arms: Treatment D
Drug: BI 44847 suspension, high dose
  Arms: Treatment A
Drug: BI 44847 tablet, low dose
  Arms: Treatment E
Drug: BI 44847 tablet, high dose
  Arms: Treatment B; Treatment C
Other: high fat breakfast
  Arms: Treatment C

SUMMARY:
Study to investigate the relative oral bioavailability of 400 mg BI 44847 as suspension vs. 400 mg BI 44847 as tablet, to investigate a food effect on the 400 mg tablet pharmacokinetic (PK) and to investigate relative oral bioavailability of 40 mg BI 44847 as solution vs. 40 mg BI 44847 as tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥ 21 and Age ≤ 50 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL) within four weeks prior to administration or during the trial
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* Any ECG value outside of the reference range and of clinical relevance including, but not limited to QRS interval > 120 ms. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 450 ms or QT> 500 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 48 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after drug administration

SECONDARY OUTCOMES:
λz (terminal rate constant in plasma) | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 48 hours after drug administration
CL/F (total clearance of the analyte in the plasma after extravascular administration) | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 48 hours after drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | up to 48 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 48 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 48 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 48 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 48 hours after drug administration
Number of patients with clinically relevant changes in vital signs | up to 3 days after last drug administration
Number of patients with clinically relevant findings in 12-lead electrocardiogram (ECG) | up to 3 days after last drug administration
Number of patients with adverse events | up to 3 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | day 3